CLINICAL TRIAL: NCT03103126
Title: The Effects of HOme-Based Combined Exercise on Glycaemic Control and Anthropometric Measurements in Patients With Type 2 Diabetes
Brief Title: HOme-Based Exercise for Patients With Type 2 Diabetes
Acronym: HOtBED
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants volunteered despite two recruitment rounds.
Sponsor: University of Portsmouth (Other)
Collaborators: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Principal Investigator, Andrew Scott, Principal Lecturer, University of Portsmouth
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HOtBED
Record Dates: First submitted 2017-03-20; First posted 2017-04-06 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: pedometer-determined walking; resistance exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Walking

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial: control group vs. one intervention arm
Who Masked: Outcomes Assessor
Masking Description: The conditions/treatments cannot be masked but the outcome assessors will be masked as to the arm that the participants are allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard care.
- Combined resistance exercise and walking (Experimental): Combined resistance exercise and walking.
  Interventions: Behavioral: Combined resistance exercise and walking

INTERVENTIONS:
Behavioral: Combined resistance exercise and walking — Combined resistance exercise and walking
  Arms: Combined resistance exercise and walking

SUMMARY:
The study aims to investigate whether 12 weeks of structured aerobic and resistance exercises completed at home can have a beneficial effect on the health of patients with type 2 diabetes compared to standard physical activity advice. The study will investigate whether the exercises can reduce factors such as patient's BMI, blood pressure and waist circumference, as well as blood glucose and insulin sensitivity. Participants will use pedometers and Therabands to carry out their exercises.

This will be compared to giving participants a physical activity advice sheet and no structured exercise examples.

DETAILED DESCRIPTION:
The study will be a 12 week randomised controlled trial, so that the researchers can isolate the independent variable of home-based combined exercise to ensure that factor is affecting the patient's measurements. Participants will be recruited from a DESMOND day through the medical team informing them of the study via a Participant Information Sheet. Once recruited and informed consent is obtained, the participants will be assigned an ID number so that they can remain anonymous, and then will be randomly allocated into either the exercise or control group. Ideally 9 participants will be recruited into each group.

All participants will be invited into the Spinnaker Physiology Laboratory at Portsmouth University at a specified date. They will have their health and fitness data collected and complete a 7-day physical activity recall questionnaire, SF-36 Form and Self-Efficacy Questionnaire before and after the intervention period to measure any change in their PA levels, self-perceived health status and self-efficacy towards exercise. They will be provided with a 7 day food diary to complete.

A control group is included so that the researchers can rule out other factors that may affect glycaemic control and anthropometric measurements. The control group will be given a Physical Activity Advice sheets as this mimics what they would normally have access to through DESMOND. The control group will receive a Physical Activity advice sheet and the researchers will talk through the advice sheet with the participants. If the control group were to have no intervention, this would be less than they normally have access to as part of their normal diabetes treatment.

The exercise group will be given the therabands and pedometer, a Physical Activity Log, Pedometer log, theraband protocol and Physical Activity Advice sheet, which will all be explained to the participant. All theraband exercises will be performed so that the researchers can ensure the participant has a good technique. The exercise intervention resistance segment will involve the exercise group performing 7 theraband exercises on three days per week on non-consecutive days. For the aerobic exercise, the participants will be asked to use the provided pedometer to record the number of steps they complete on day 1 of the intervention (assuming that on this day, they complete their normal daily activities that they would do most days of the week). They then are asked to add 2,000 steps onto their daily steps; this amount will then become their daily step goal. Once they have reached this goal on 4 out of 5 days, they are asked to increase their step goal by 500.

The participants will be invited back after 12 weeks to repeat the pre-study measures to assess any changes.

ELIGIBILITY:
Inclusion Criteria:

* Participants must not be meeting the government's recommended physical activity guideline (150 min moderate intensity exercise per week)
* Must be 18 years of age or over
* Diagnosed with Type 2 Diabetes and have been referred to DESMOND, as this is where they will be recruited from.

Exclusion Criteria:

● Co-morbidity that prevents them undertaking physical activity safely, such as cardiac disease or pulmonary disease or significant musculoskeletal limitations. This will be determined from the Exercise and Health History Questionnaire. If their diabetes is severe and they have peripheral neuropathy or any associated systemic, cardiovascular, metabolic or musculoskeletal problems which will inhibit their ability to perform exercise safely.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender is not an eligibility or outcome measure so self-representation will suffice as an indicator
Enrollment: 0 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
The effects of home-based combined exercise on insulin sensitivity compared to physical activity advice during the 6 week study period | 6 weeks
  Insulin sensitivity will be calculated from plasma glucose and serum insulin measures

SECONDARY OUTCOMES:
The effects of HBCE on body mass index (BMI) compared to physical activity advice during the 6 week study period | 6 weeks
  Height and body mass will be measured to determine whether the intervention improves BMI (kg.m2)
The effects of HBCE on waist circumference compared to physical activity advice during the 6 week study period | 6 weeks
  To determine whether the intervention improves waist circumference in centimetres
The effects of HBCE on body fat percentage compared to physical activity advice during the 6 week study period | 6 weeks
  To determine whether the intervention improves body fat percentage using bioelectrical impedance analysis
The effect of HBCE on physical activity levels compared to physical activity advice during the 6 week study period | 6 weeks
  To determine if HBCE is more effective at increasing physical activity compared to physical activity advice using an International Physical Activity Questionnaire at baseline and the last week of the study period.
The effect of HBCE on fitness compared to physical activity advice during the 6 week study period | 6 weeks
  To determine if HBCE is more effective at increasing fitness levels compared to physical activity advice using the Tecumseh step test, a modified version of the Harvard step test (Shorter test period and shorter step).
The number of participants recruited and the average number per week | 6 weeks
  Can sufficient participant numbers can be recruited from a DESMOND day? The number of participants recruited and average per week of recruitment will be recorded and calculated.
The percentage adherence to the home-based combined exercise programme | 6 weeks
  Adherence to the home-based combined exercise programme will be monitored in a diary
Self-perceived health status measured using the SF-36 quality of life scale | 6 weeks
  The SF36 will be applied at baseline and post-intervention in both groups to determine any changes and differences between control vs exercise groups
Self-efficacy to regulate exercise scale | 6 weeks
  The self-efficacy to regulate exercise scale will be applied at baseline and post-intervention in both groups to determine any changes and differences between control vs exercise groups

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T Scott, PhD, Study Chair — University of Portsmouth
Locations (1):
- Andrew Scott, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The data will be stored in link-anonymised form and will not be made available outside of the research team.